CLINICAL TRIAL: NCT06706492
Title: Comparison of Muscle Oxygenation, Functional Capacity, and Frailty in Kidney Transplant Recipients with and Without Inspiratory Muscle Weakness
Brief Title: Muscle Oxygenation, Functional Capacity and Frailty in Kidney Transplant Recipients with and Without Inspiratory Muscle Weakness
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: SBA 23/286
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with inspiratory muscle weakness
- Patients without inspiratory muscle weakness

SUMMARY:
The aim of this study was to compare respiratory function, muscle oxygenation, functional capacity, peripheral muscle strength, body composition, and frailty in kidney transplant recipients with and without inspiratory muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney transplantation
* At least 6 months after the kidney transplant
* Not having regular exercise habits
* Voluntary participation in the study

Exclusion Criteria:

* Having a musculoskeletal problem that may interfere with the tests
* Having neurological impairment
* Having chronic lung disease
* Having had any cardiovascular event in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | 1st day
  Maximal inspiratory pressure (MIP) will be measured using a portable mouth pressure measuring device.
Respiratory muscle strength | 1st day
  Maximal expiratory pressure (MEP) will be measured using a portable mouth pressure measuring device.
Functional capacity | 1st day
  Will be evaluated with 6 minute walk test.
Peripheral muscle strength | 1st day
  Knee extensor strength will be measured using a hand dynamometer.
Peripheral muscle strength | 1st day
  Hand grip strength will be measured using grip dynamometer.

SECONDARY OUTCOMES:
Forced expiratory volume in one second | 1st day
  Respiratory function will be evaluated using spirometry. Forced expiratory volume in one second will be recorded.
Forced vital capacity | 1st day
  Respiratory function will be evaluated using spirometry. Forced vital capacity will be recorded.
Forced expiratory volume in one second/forced vital capacity | 1st day
  Respiratory function will be evaluated using spirometry. Forced expiratory volume in one second/forced vital capacity will be recorded.
Peak expiratory flow | 1st day
  Respiratory function will be evaluated using spirometry. Peak expiratory flow will be recorded.
Forced mid-expiratory flow | 1st day
  Respiratory function will be evaluated using spirometry. Forced mid-expiratory flow (FEF25-75) will be recorded.
Body composition | 1st day
  It will be evaluated by bioelectrical impedance analysis method. Percentage of fat and lean body mass wiil be recorded.
Fragility | 1st day
  It will be assessed according to the criteria defined by Fried. The existence of 5 parameters is questioned here. These parameters are as follows: weight loss, weakness, fatigue, slowness, low physical activity. Those with 3 or more of the 5 identified components are classified as fragile.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)